CLINICAL TRIAL: NCT07333378
Title: Post-partum Retention of Vernix Caseosa for Primary Prevention of Atopic Dermatitis, Guarding Skin Integrity and Fostering a Healthy Microbiome.
Brief Title: Retention of Vernix Caseosa in Newborns for Primary Prevention of Atopic Dermatitis
Acronym: PROTEGO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 230610001; 1241933 (Other Grant/Funding Number: Agencia Nacional de Investigación y Desarrollo / FONDECYT (Chile))
Record Dates: First submitted 2025-12-05; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
Keywords: vernix caseosa; primary prevention; newborn; eczema; atopic dermatitis; skin infections; Staphylococcus aureus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Cellulitis; Staphylococcal Infections

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, controlled, parallel-group trial conducted in three maternity hospitals in Santiago, Chile. Mother-infant pairs are assigned 1:1 to either vernix retention (experimental) or vernix removal (control). In the retention arm, vernix caseosa is left on the skin and bathing is delayed ≥24 h; in the control arm, vernix is removed within 2 hours per standard care. Randomization is centralized via an Interactive Response Technology (IRT) system and stratified by site, delivery mode, and parental atopy. The study uses a single-blind (assessor-blinded) design with 12-month follow-up. Primary purpose: prevention of atopic dermatitis through improved skin-barrier and microbiome development.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, masking of mothers, families, and delivery staff is not feasible. The trial uses a single-blind design, where outcome assessors, investigators performing clinical evaluations, data analysts, and laboratory personnel are blinded to treatment allocation. Randomization and group assignment are managed centrally through a secure Interactive Response Technology (IRT) system to ensure allocation concealment. Study documentation and sample labels use coded identifiers to maintain blinding throughout data collection and analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retain vernix caseosa (Experimental): After delivery, visible blood and fluids are gently wiped from the newborn's skin while leaving the vernix caseosa intact. Bathing or cleansing with water or oil is delayed for at least 24 hours (preferably up to 7 days) according to the study protocol. Excess vernix may be lightly spread across the body surface to ensure even coverage. Standard thermal care, skin-to-skin contact, and other routine newborn procedures are maintained. No emollients or cleansers are applied during the retention period.
  Interventions: Other: Retention of Vernix Caseosa After Birth
- Early removal of vernix caseosa (Other): Within two hours after birth, newborns receive standard hospital cleansing with sterile water and vegetable oil or petroleum jelly to completely remove vernix caseosa, blood, and other residues. The procedure follows routine postnatal care practices at each participating site. After cleaning, usual thermal care, dressing, and parental skin-to-skin contact are continued. No experimental procedures or restrictions are applied beyond standard care.
  Interventions: Other: Removal of Vernix Caseosa After Birth

INTERVENTIONS:
Other: Retention of Vernix Caseosa After Birth — Retention of vernix caseosa on the newborn's skin after birth by avoiding early cleaning or bathing for ≥24 hours, allowing it to dry and absorb naturally.
  Arms: Retain vernix caseosa
Other: Removal of Vernix Caseosa After Birth — Early removal of vernix caseosa from the newborn's skin within the first two hours after birth by washing the child with water and petroleum jelly or vegetable oil, as is standard practice in study hospitals.
  Arms: Early removal of vernix caseosa

SUMMARY:
Atopic dermatitis (AD), also known as eczema, is a common chronic inflammatory skin disease that usually begins in infancy and causes significant itching, discomfort, and sleep disturbance. It affects up to one in five children worldwide and represents a growing public-health problem. Research has shown that genetic and environmental factors contribute to its development, especially those related to skin-barrier integrity and the skin microbiome during early life. Preventing AD before it starts-known as primary prevention-has become an important goal.

Vernix caseosa is a naturally occurring, white, creamy substance that covers the skin of newborns at birth. It forms during the last trimester of pregnancy and plays a key role in protecting and hydrating the baby's skin before and after birth. Vernix contains water, lipids, and proteins with antimicrobial and anti-inflammatory properties. Despite these potential benefits, in many hospitals vernix is routinely removed soon after delivery as part of standard newborn cleaning or bathing practices. However, there is little scientific evidence to support early removal, and some studies suggest that keeping vernix on the skin for longer may help the newborn's skin barrier function and reduce colonization by harmful bacteria.

The PROTEGO Study (Post-Partum Retention of Vernix Caseosa for Primary Prevention of Atopic Dermatitis, Guarding Skin Integrity and Fostering a Healthy Microbiome) is a randomized controlled clinical trial designed to test whether delaying the removal of vernix caseosa after birth can help prevent atopic dermatitis and improve skin health during the first year of life.

A total of 1,383 mother-infant pairs will be enrolled from three maternity hospitals in Santiago, Chile. Participants will be randomly assigned to one of two groups:

1. Retention group: Vernix caseosa will be left on the skin and allowed to dry naturally; the baby's first bath will be delayed according to the study protocol.
2. Removal group: Vernix will be removed following current hospital practice using gentle cleaning with water and oil or petroleum jelly shortly after birth.

All infants will be followed for 12 months with regular clinical assessments, standardized skin evaluations, and collection of biological samples. The main outcome will be the cumulative incidence of atopic dermatitis, diagnosed using modified UK Working Party criteria and/or Hanifin & Rajka criteria at 12 months of age. Secondary outcomes include skin-barrier measurements (transepidermal water loss, skin pH, and natural moisturizing factor), the composition of the skin microbiome, and early signs of allergic or infectious diseases.

This study will provide high-quality evidence on whether preserving vernix caseosa after birth is a simple, safe, cost-effective and natural strategy to strengthen the newborn's skin barrier and reduce the risk of eczema and related conditions. The results could help improve newborn-care practices and promote skin health in early life worldwide.

DETAILED DESCRIPTION:
Scientific Rationale:

Atopic dermatitis (AD) is a chronic, relapsing, inflammatory skin disorder that typically begins in early childhood and is characterized by pruritic eczematous lesions, epidermal barrier dysfunction, and immune dysregulation. Its prevalence is rising globally, affecting 10-35 % of children in industrialized countries. In Chile, epidemiological studies show that 18-22 % of school-aged children and up to one third of toddlers have physician-diagnosed AD, indicating a substantial and increasing disease burden. AD is often the first manifestation of the "atopic march," leading to food allergy, asthma, and allergic rhinitis.

Although several biologic and small-molecule therapies have recently transformed the management of moderate-to-severe AD, these treatments remain costly, inaccessible for most patients, and do not prevent disease onset. Therefore, identifying effective and feasible primary prevention strategies is a major unmet need.

Current understanding of AD pathogenesis highlights three interacting domains: (1) structural and biochemical defects of the epidermal barrier; (2) skewed type-2 immune responses; and (3) altered skin microbiota with increased colonization by Staphylococcus aureus. Defects in epidermal proteins such as filaggrin (FLG) increase transepidermal water loss (TEWL) and permeability to allergens and microbes, while immune activation and microbial imbalance perpetuate inflammation. Because these abnormalities emerge early in life-often before clinical symptoms-interventions targeting skin-barrier maturation and microbial balance during the neonatal period may reduce AD incidence.

Vernix Caseosa as a Natural Barrier Protector:

Vernix caseosa (VC) is a unique biofilm-like substance produced in utero by fetal sebaceous glands and composed of water (≈ 80 %), lipids (≈ 10 %), and proteins (≈ 10 %) intermingled with corneocytes. It covers the fetus during the third trimester, protecting the skin from maceration in the amniotic environment and promoting terminal differentiation of the stratum corneum. VC exhibits semipermeable and antimicrobial properties, functioning as a physiological barrier and innate immune interface. Its lipids include ceramides, cholesterol, and free fatty acids-key constituents of postnatal epidermal barrier repair-while its proteins include antimicrobial peptides such as LL-37, psoriasin, RNase 7, and lysozyme, as well as enzymes involved in lipid metabolism.

Despite these potential benefits, in many institutions worldwide VC is routinely removed within hours after birth as part of standard newborn cleaning procedures. Early removal eliminates a biologically active matrix that may support optimal skin barrier transition from intrauterine to extrauterine life. Small randomized and observational studies suggest that delaying vernix removal increases skin hydration, lowers skin pH, and may reduce bacterial colonization by S. aureus and E. coli, but evidence is limited by short follow-up and small sample sizes and no studies have evaluated its long-term impact on incidence of atopic dermatitis and other conditions.

The PROTEGO trial aims to test whether retaining vernix caseosa after birth, compared with its routine early removal, reduces the risk of developing AD during the first year of life and improves biophysical and microbiological indicators of skin health.

Study Design:

PROTEGO is a multicenter, randomized, controlled, parallel-group clinical trial with assessor blinding. The trial will enroll 1,383 pregnant women and their newborns from three high-volume maternity hospitals in Santiago, Chile. Eligible participants are healthy mothers ≥ 18 years of age with singleton pregnancies and expected delivery of a healthy neonate (≥ 34 weeks, birthweight ≥ 2000 g). After written informed consent, participants will be randomly assigned 1:1 via a centralized interactive response technology (IRT) system to either the vernix retention group or the vernix removal group. Randomization is stratified by clinical site, mode of delivery (vaginal/cesarean), and parental history of atopy.

Because masking of the delivery team and parents is not feasible, the study will use single-blind assessment, ensuring that investigators evaluating outcomes remain unaware of group assignment. Participants will be followed from birth to 12 months through scheduled visits (at 24-96 h; 7 days; and 1, 3, 6, 9, and 12 months).

Safety and Monitoring:

Retention or removal of VC are standard practices varying between institutions and are considered a minimal-risk intervention. Potential risks include mild skin irritation, transient erythema, or theoretical risk of hypothermia if bathing is delayed excessively. These will be mitigated by standard neonatal thermal-care protocols and skin monitoring. Adverse events (AEs) and serious adverse events (SAEs) will be actively monitored and reported according to institutional and national regulations.

Expected Impact:

If vernix retention proves effective, this trial could introduce a simple, low-cost, and universally applicable strategy for the primary prevention of atopic dermatitis. Because the intervention involves modifying routine newborn care rather than introducing new drugs or devices, it has high translational potential for maternity wards worldwide, especially in low- and middle-income settings.

Beyond its clinical endpoint, PROTEGO will generate valuable mechanistic insights into early-life skin-barrier biology, the neonatal microbiome, and gene-environment interactions (e.g., FLG variants). The integrated biophysical, microbiological, and transcriptomic datasets may illuminate new pathways linking perinatal skin care and immune development. PROTEGO is the first large-scale randomized controlled trial evaluating whether the simple act of preserving vernix caseosa after birth can prevent atopic dermatitis. By combining clinical follow-up with state-of-the-art barrier and microbiome analyses, this study seeks to redefine evidence-based newborn-skin care and contribute to global efforts to reduce the burden of allergic and inflammatory diseases from the very beginning of life.

ELIGIBILITY:
Inclusion Criteria:

* pregnant mother aged 18 and older, who is able to provide informed consent for participation
* delivery of a healthy, singleton newborn (vaginal or cesarean) at one of the study sites.
* parents are able and willing to comply with the study schedule and procedures

Exclusion Criteria:

* birthweight <2000 g
* prematurity younger than 34 weeks of gestation
* multiple gestation / multiple births
* maternal HIV-positivity
* clinical and/or laboratory diagnosis of chorioamnionitis.
* need for neonatal hospitalization or presence of an acute illness (e.g., neonatal respiratory distress syndrome) within the first 24 hours of life.
* severe and generalized congenital skin disorder (e.g., congenital ichthyosis).

Min Age: 0 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1383 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of atopic dermatitis at 1 year of age | 12 months
  Proportion of infants who meet the diagnostic criteria for atopic dermatitis at 12 months of age, assessed using the modified UK Working Party criteria and/or Hanifin & Rajka criteria, evaluated by a trained assessor blinded to group allocation.

SECONDARY OUTCOMES:
Incidence of Atopic Dermatitis (Hanifin & Rajka Criteria Only) | 12 months.
  Proportion of infants diagnosed with atopic dermatitis at 12 months using only the Hanifin & Rajka criteria.
Cumulative Incidence of Atopic Dermatitis (Modified UK Working Party Criteria Only) | 0-12 months
  Proportion of infants diagnosed with atopic dermatitis using only the modified UK Working Party criteria for atopic dermatitis at any study contact until 12 months.
Cumulative Incidence of Infant Eczema | 0-12 months
  Proportion of infants with any eczema skin lesions (clinician or parent-reported) up to 12 months of age.
Atopic dermatitis diagnosed by trained physician | 12 months
  Diagnosis of atopic dermatitis by a trained physician using standard clinical criteria at 12 months of age
Parent-reported atopic dermatitis | 0-12 months
  Parental report of a physician diagnosis of atopic dermatitis collected via standardized questionnaire.
Cumulative incidence of atopic dermatitis by CEQ at 12 months | 0-12 months
  Cumulative incidence of AD diagnosed using the Children's Eczema Questionnaire (CEQ).
Use of topical anti-inflammatory medications | 0-12 months
  Any reported use of atopic dermatitis topical medications, such as corticosteroids or calcineurin inhibitors, during the first 12 months of age.
Time to onset of AD based on parent-reported age at first appearance among infants with AD | From birth to 12 months of age
  Time to onset of AD based on parent-reported age at first appearance among infants with AD.
AD severity measured by the Patient-Oriented Eczema Measure (POEM) among infants with AD | From birth to 12 months of age
  AD severity measured by the Patient-Oriented Eczema Measure (POEM) among infants with AD.
Severity of Atopic Dermatitis (SCORAD) among infants with AD | 12 months of age
  Severity of Atopic Dermatitis (SCORAD) among infants with AD at 12 months of age.
Global AD severity based on parental assessment among infants with AD | From birth to 12 months of age
  Global AD severity based on parental assessment among infants with AD.
Interaction of intervention with visible vernix caseosa (VC) at birth | 0-12 months
  Evaluate the effects of the amount of visible VC on the incidence of AD in the intervention and control groups.
Interaction of intervention with FLG loss-of-function mutations | 0-12 months
  Evaluate the effects of FLG loss-of-function mutations on the incidence of AD in the intervention and control groups.
Dynamics of Staphylococcal Colonization | 0-12 months
  Cumulative incidence of positive Staphylococcus aureus (and other Staphylococcal species) identification on the skin during the first year of life.
Transepidermal water loss (TEWL) at 24-96 hours of age | 24-96 hours
  Measurement of transepidermal water loss (TEWL) at 24-96 hours of age
Transepidermal water loss (TEWL) at 12 months of age | 12 months of age
  Measurement of transepidermal water loss (TEWL) at 12 months of age.
Skin pH at 24-96 hours of age | 24-96 hours of age
  Measurement of skin pH at 24-96 hours of age.
Skin pH at 12 months of age | 12 months of age
  Measurement of skin pH at 12 months of age.
Epidermal natural moisturizing factor (NMF) concentration at 12 months. | 12 months of age
  Epidermal natural moisturizing factor (NMF) concentration in tape stripping samples at 12 months of age.

OTHER OUTCOMES:
Newborn temperature regulation | 0-24 hours of life
  Serial measurements of body temperature during the first 24 hours of life.
Serious bacterial infections | 28 and 90 days of life
  Incidence of serious bacterial infections at 28 and 90 days.
Skin infections during infancy | 0-12 months
  Cumulative incidence of bacterial skin infections during the first 12 months of life.
Parent-reported food allergy incidence | 12 months
  Cumulative incidence of food allergy based on Parent-reported immediate symptoms of food allergy.
Physician-diagnosed food allergy incidence | 12 months
  Cumulative incidence of food allergy based on parent-reported physician-diagnosed food allergy confirmed by skin-prick test, specific IgE, or oral food challenge.
Parental Acceptability of Vernix Retention vs. Removal | 12 months
  Acceptability and satisfaction with assigned intervention assessed via parental questionnaire.
Type-2 immunity biomarkers in stratum corneum transcriptomics | 12 months of age
  Comparison of gene-expression markers of type-2 immunity in the stratum corneum at 12 months between VC retention and early removal groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Clínica San Carlos de Apoquindo, Las Condes, RM
  - Hospital Clínico Universidad Católica, Santiago, RM

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be shared upon reasonable request.

REFERENCES:
- [Background] Endre KMA, Landro L, LeBlanc M, Gjersvik P, Lodrup Carlsen KC, Haugen G, Hedlin G, Jonassen CM, Nordlund B, Rudi K, Skjerven HO, Staff AC, Soderhall C, Vettukattil R, Rehbinder EM. Diagnosing atopic dermatitis in infancy using established diagnostic criteria: a cohort study. Br J Dermatol. 2022 Jan;186(1):50-58. doi: 10.1111/bjd.19831. Epub 2021 May 6. PMID 33511639
- [Background] Tejos-Bravo M, Venegas L, Iturriaga C, Sabatini N, Martin C, Pérez-Mateluna G, Urzúa M, Cabalín C, Dossi MT, Del Barrio P, Majerson D, Silva-Valenzuela S, Vera-Kellet C, Borzutzky A. Alterations in skin physiology are associated with disease severity in Chilean patients with atopic dermatitis. European Academy of Allergy and Immunology Congress 2019. Lisbon, Portugal. June 1-5, 2019.
- [Background] Ahmed SOM. Vernix Caseosa: Benefits and Clinical Implications in Neonatal Care;A Study Conducted at Almak Nimr University Hospital, Shendi, Sudan. Int J Environ Sci. 2025; 11(469-475).
- [Background] Blume-Peytavi U, Cork MJ, Faergemann J, Szczapa J, Vanaclocha F, Gelmetti C. Bathing and cleansing in newborns from day 1 to first year of life: recommendations from a European round table meeting. J Eur Acad Dermatol Venereol. 2009 Jul;23(7):751-9. doi: 10.1111/j.1468-3083.2009.03140.x. PMID 19646134
- [Background] Wisniewski JA, Phillipi CA, Goyal N, Smith A, Hoyt AEW, King E, West D, Golden WC, Kellams A. Variation in Newborn Skincare Policies Across United States Maternity Hospitals. Hosp Pediatr. 2021 Sep;11(9):1010-1019. doi: 10.1542/hpeds.2021-005948. PMID 34462323
- [Background] Henningsson A, Nystrom B, Tunnell R. Bathing or washing babies after birth? Lancet. 1981 Dec 19-26;2(8260-61):1401-3. doi: 10.1016/s0140-6736(81)92812-9. PMID 6118769
- [Background] Bergstrom A, Byaruhanga R, Okong P. The impact of newborn bathing on the prevalence of neonatal hypothermia in Uganda: a randomized, controlled trial. Acta Paediatr. 2005 Oct;94(10):1462-7. doi: 10.1111/j.1651-2227.2005.tb01821.x. PMID 16299878
- [Background] Jha AK, Baliga S, Kumar HH, Rangnekar A, Baliga BS. Is There a Preventive Role for Vernix Caseosa?: An Invitro Study. J Clin Diagn Res. 2015 Nov;9(11):SC13-6. doi: 10.7860/JCDR/2015/14740.6784. Epub 2015 Nov 1. PMID 26674069
- [Background] Cabalin C, Dibarrart M, Nunez-Rosales JJ, Faunes M, Avaca M, Avalos P, Fabres J, Alvarez-Figueroa MJ, Vera-Kellet C, Silva-Valenzuela S, Saez CG, Borzutzky A. Vernix caseosa reveals mechanistic clues linking maternal obesity to atopic dermatitis pathogenesis. J Allergy Clin Immunol. 2024 Mar;153(3):860-867.e1. doi: 10.1016/j.jaci.2023.09.042. Epub 2023 Dec 2. PMID 38048884
- [Background] Akinbi HT, Narendran V, Pass AK, Markart P, Hoath SB. Host defense proteins in vernix caseosa and amniotic fluid. Am J Obstet Gynecol. 2004 Dec;191(6):2090-6. doi: 10.1016/j.ajog.2004.05.002. PMID 15592296
- [Background] Yoshio H, Tollin M, Gudmundsson GH, Lagercrantz H, Jornvall H, Marchini G, Agerberth B. Antimicrobial polypeptides of human vernix caseosa and amniotic fluid: implications for newborn innate defense. Pediatr Res. 2003 Feb;53(2):211-6. doi: 10.1203/01.PDR.0000047471.47777.B0. PMID 12538777
- [Background] Marchini G, Lindow S, Brismar H, Stabi B, Berggren V, Ulfgren AK, Lonne-Rahm S, Agerberth B, Gudmundsson GH. The newborn infant is protected by an innate antimicrobial barrier: peptide antibiotics are present in the skin and vernix caseosa. Br J Dermatol. 2002 Dec;147(6):1127-34. doi: 10.1046/j.1365-2133.2002.05014.x. PMID 12452861
- [Background] Holm T, Rutishauser D, Kai-Larsen Y, Lyutvinskiy Y, Stenius F, Zubarev RA, Agerberth B, Alm J, Scheynius A. Protein biomarkers in vernix with potential to predict the development of atopic eczema in early childhood. Allergy. 2014 Jan;69(1):104-12. doi: 10.1111/all.12308. Epub 2013 Nov 11. PMID 24205894
- [Background] Tollin M, Jagerbrink T, Haraldsson A, Agerberth B, Jornvall H. Proteome analysis of vernix caseosa. Pediatr Res. 2006 Oct;60(4):430-4. doi: 10.1203/01.pdr.0000238253.51224.d7. Epub 2006 Aug 28. PMID 16940245
- [Background] Svendsen EK, Grundt I. Total lipids and lipid pattern in amniotic fluid and vernix caseosa. A preliminary report. Acta Obstet Gynecol Scand. 1966;45(S9):80-3. doi: 10.3109/00016346609158604. No abstract available. PMID 5958408
- [Background] Biezenski JJ, Pomerance W, Goodman J. Studies on the origin of amniotic fluid lipids. I. Normal composition. Am J Obstet Gynecol. 1968 Nov 15;102(6):853-61. doi: 10.1016/0002-9378(68)90514-0. No abstract available. PMID 5686904
- [Background] Wysocki SJ, Grauaug A, O'Neill G, Hahnel R. Lipids in forehead vernix from newborn infants. Biol Neonate. 1981;39(5-6):300-4. doi: 10.1159/000241452. PMID 7260215
- [Background] Tollin M, Bergsson G, Kai-Larsen Y, Lengqvist J, Sjovall J, Griffiths W, Skuladottir GV, Haraldsson A, Jornvall H, Gudmundsson GH, Agerberth B. Vernix caseosa as a multi-component defence system based on polypeptides, lipids and their interactions. Cell Mol Life Sci. 2005 Oct;62(19-20):2390-9. doi: 10.1007/s00018-005-5260-7. PMID 16179970
- [Background] Rissmann R, Groenink HW, Weerheim AM, Hoath SB, Ponec M, Bouwstra JA. New insights into ultrastructure, lipid composition and organization of vernix caseosa. J Invest Dermatol. 2006 Aug;126(8):1823-33. doi: 10.1038/sj.jid.5700305. Epub 2006 Apr 20. PMID 16628195
- [Background] Mikova R, Vrkoslav V, Hanus R, Hakova E, Habova Z, Dolezal A, Plavka R, Coufal P, Cvacka J. Newborn boys and girls differ in the lipid composition of vernix caseosa. PLoS One. 2014 Jun 9;9(6):e99173. doi: 10.1371/journal.pone.0099173. eCollection 2014. PMID 24911066
- [Background] Checa A, Holm T, Sjodin MO, Reinke SN, Alm J, Scheynius A, Wheelock CE. Lipid mediator profile in vernix caseosa reflects skin barrier development. Sci Rep. 2015 Nov 2;5:15740. doi: 10.1038/srep15740. PMID 26521946
- [Background] Oudshoorn MH, Rissmann R, van der Coelen D, Hennink WE, Ponec M, Bouwstra JA. Development of a murine model to evaluate the effect of vernix caseosa on skin barrier recovery. Exp Dermatol. 2009 Feb;18(2):178-84. doi: 10.1111/j.1600-0625.2008.00780.x. Epub 2008 Aug 4. PMID 18684123
- [Background] Bautista MI, Wickett RR, Visscher MO, Pickens WL, Hoath SB. Characterization of vernix caseosa as a natural biofilm: comparison to standard oil-based ointments. Pediatr Dermatol. 2000 Jul-Aug;17(4):253-60. doi: 10.1046/j.1525-1470.2000.01770.x. PMID 10990571
- [Background] Pickens WL, Warner RR, Boissy YL, Boissy RE, Hoath SB. Characterization of vernix caseosa: water content, morphology, and elemental analysis. J Invest Dermatol. 2000 Nov;115(5):875-81. doi: 10.1046/j.1523-1747.2000.00134.x. PMID 11069626
- [Background] Hoeger PH, Schreiner V, Klaassen IA, Enzmann CC, Friedrichs K, Bleck O. Epidermal barrier lipids in human vernix caseosa: corresponding ceramide pattern in vernix and fetal skin. Br J Dermatol. 2002 Feb;146(2):194-201. doi: 10.1046/j.1365-2133.2002.04584.x. PMID 11903227
- [Background] Visscher MO, Narendran V, Pickens WL, LaRuffa AA, Meinzen-Derr J, Allen K, Hoath SB. Vernix caseosa in neonatal adaptation. J Perinatol. 2005 Jul;25(7):440-6. doi: 10.1038/sj.jp.7211305. PMID 15830002
- [Background] Visscher MO, Barai N, LaRuffa AA, Pickens WL, Narendran V, Hoath SB. Epidermal barrier treatments based on vernix caseosa. Skin Pharmacol Physiol. 2011;24(6):322-9. doi: 10.1159/000328744. Epub 2011 Aug 4. PMID 21822033
- [Background] Cardenas GV, Iturriaga C, Hernandez CD, Tejos-Bravo M, Perez-Mateluna G, Cabalin C, Urzua M, Venegas-Salas LF, Fraga JP, Rebolledo B, Poli MC, Repetto GM, Casanello P, Castro-Rodriguez JA, Borzutzky A. Prevalence of filaggrin loss-of-function variants in Chilean population with and without atopic dermatitis. Int J Dermatol. 2022 Mar;61(3):310-315. doi: 10.1111/ijd.15887. Epub 2021 Sep 4. PMID 34480753
- [Background] Borzutzky A, Cabalin C. From Thin to Thick: Weight Gain in Children Feeds the Risk of Atopic Dermatitis. J Invest Dermatol. 2024 Sep;144(9):1909-1911. doi: 10.1016/j.jid.2024.02.035. Epub 2024 May 14. No abstract available. PMID 38752941